CLINICAL TRIAL: NCT03968666
Title: Evaluation of Compliance With Enhanced Recovery After Surgery (ERAS) Protocol in Benign Gynecological Surgical Patients
Brief Title: Compliance With Enhanced Recovery After Surgery Protocol (ERAS) in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor, Augusta University
Other Study IDs: 1396793
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Surgery; Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecological surgery with ERAS protocol: Patients scheduled for benign gynecological surgery under ERAS protocol

SUMMARY:
The concept of "enhanced recovery" was introduced by European anesthesiologists and surgeons who challenged traditional clinical practices involved in peri-operative care in 1990s. The goal of enhanced recovery programs (ERP) is to maintain normal physiology thereby decreasing complications. It focuses on peri-operative optimization of patient care. It was originally created for open colorectal surgeries but now has shown benefit in various surgical specialities including thoracic surgery, vascular surgery, hepatobiliary as well as gynecological surgery.

The successful implementation of structured ERAS program requires an ERAS protocol, audit system and a multidisciplinary team. The investigators will evaluate the effect of compliance with the protocol and outcomes such as length of stay, readmissions, morbidity and mortality.

DETAILED DESCRIPTION:
After approval by the Institutional Review Board, the investigators plan to retrospectively study gynecological patients who underwent ERAS protocol at Augusta University Medical Center between January 2017 and February 2019.

This is a retrospective observational study to evaluate the outcomes of patients who had ERAS protocol during their surgery.

Demographic and outcome variables will be obtained from the institutional health documentation system. The investigators will collect demographic variables (age, ASA status), morphometric measurements (body mass index), time from enrollment to ERAS protocol, hospitalization length of stay, and readmission rate. The investigators will also record the documentation of the ERAS protocol interventions against the ERAS protocol approved by the institution. The investigators will assess the effect of the degree of compliance on outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* All elective benign gynecological surgical patients enrolled under ERAS protocol

Exclusion Criteria:

* History of oncologic pathologies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecological surgery
Study Population: Patients scheduled for benign gynecologic surgery who underwent ERAS protocol
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay | 2 weeks
  Days from surgery to discharge from the hospital

SECONDARY OUTCOMES:
Readmission | 2 weeks
  Admission to hospital after discharge
Mortality | 2 weeks
  Number of fatalities after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros Perez, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided